CLINICAL TRIAL: NCT03516448
Title: Randomized, Double-Blind, Placebo-Controlled, Multicenter Expanding Phase III Clinical Trial to Evaluate the Safety and Efficacy of Injectable Tyroserleutide to Treat Hepatocellular Carcinoma (HCC) (After HCC Resection)
Brief Title: Expanding Phase III Study of Tyroserleutide for Injection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shenzhen Kangzhe Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TYS-CN-1.1PUMP III(C)
Record Dates: First submitted 2017-07-04; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — H-Tyr-Ser-Leu-OH; Injections

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Tyroserleutide for injection (Active Comparator): the Tyroserleutide for injection at the dosage of 6mg/d Gan Fu Le Tablets，6 tablets,po,tid
  Interventions: Drug: Gan Fu Le Tablets; Drug: Tyroserleutide for injection
- the placebo group (Placebo Comparator): the placebo Gan Fu Le Tablets，6 tablets,po,tid
  Interventions: Drug: Gan Fu Le Tablets; Drug: Placebo

INTERVENTIONS:
Drug: Gan Fu Le Tablets — 6 Tablets，tid,po
Drug: Tyroserleutide for injection — 6mg/d, 5days,ivgtt
  Arms: the Tyroserleutide for injection
Drug: Placebo — 0mg/d, 5days,ivgtt
  Arms: the placebo group

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, multi-center Clinical Trial. Patients with no tumor lesions 21 days after resection of hepatocellular carcinoma will be randomized in a 1:1 ratio to 1 of the 2 treatment groups：6mg/d Tyroserleutide (injection), or placebo

DETAILED DESCRIPTION:
* The first stage includes evaluation of subjects, to assess the inclusion criteria and exclusion criteria, based on the patients' preoperative imaging results, including tumor size, tumor characteristics, etc.
* In the second stage, subjects will return to the hospital 21 days following the baseline examination.The investigator will determine whether the subject satisfies all inclusion/exclusion criteria. If all requirements are satisfied, then randomization will occur 21 days after surgery
* The day of randomization will be defined as Day 0. Randomized subjects will return to the hospital and begin cycle 1 on the day of randomization (Day 0). and the relevant laboratory tests will be performed within 3 days after the end the study drug infusion.
* Cycles will occur as follows: cycles 2, 3, 4, 5, and n will begin on days 42±3, 70±3, 98±3, 126±3, and 14+28（n-1)± 3, respectively.
* Based therapeutic drugs are Gan Fu Le
* the participant will receive medical inspection so as to observe and ensure drug safety.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Aged ≥ 18 years and ≤ 75 years old, male or female
* Subject underwent resection of hepatocellular carcinoma (confirmed by pathology)
* The tumor characteristics must meet the following:A single tumor with a maximum diameter >5cm ,Preoperative imaging, or Intraoperative visual observation.;

Exclusion Criteria:

* Concomitant malignant tumor(s) in other systems is/are present
* Tumor thrombosis in the branch of portal vein or in hepatic vein is detected by preoperative imaging or observed during the surgery
* The subject received any previous systemic anti-HCC therapy prior to the resection surgery (except the resection surgery), such as liver transplantation, intervention, ablation, radiotherapy, chemotherapy, molecular targeted therapy or other anti-HCC therapy
* The subject took Sorafenib prior to randomization
* The subject took other study/investigational drugs 7 days prior to randomization
* The subject took Kang Laike injection/soft capsule，or Jinke Huaier granule 7 days prior to randomization
* The subject has central nervous system disease, mental illness, unstable angina, congestive heart failure, severe arrhythmia or other severe uncontrolled diseases
* The subject has history of investigational drug or similar drug allergy
* The baseline examination indicates that infection, bleeding, bile leakage, or other postoperative complications are present
* The subject is pregnant, lactating, or urine pregnancy test result is positive
* Baseline (post-resection) examination exist tumor recurrence or metastasis;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2016-06-13 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
OS （Overall Survival） | 3 years
  The time from randomization to death due to any reason

SECONDARY OUTCOMES:
RFS(Recurrence Free Survival) | 3 years
  The time from randomization to recurrence, metastasis or death due to any reason